CLINICAL TRIAL: NCT01272765
Title: Surveillance Study of Weight Response and Body Composition in Subjects Taking a Stable Dose of Risperdal, Seroquel, and/or Zyprexa for Greater Than 3 Months in Combination With 500 mg IHBG-10 TID
Brief Title: Anti-psychotic Medication (Stable Dose) Weight Loss Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study did not get started.
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARI-1320-IHBG10
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Obesity
Keywords: obesity; weight loss; weight management; anti-psychotic medication; Zyprexa; Seroquel; Risperdal
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control Group (Placebo Comparator)
  Interventions: Other: Placebo
- Risperdal Group (Experimental): Subjects who are on a stable dose of Ripserdal and taking 500 mg IHBG-10 15 minutes prior to the three main meals of the day.
  Interventions: Dietary Supplement: IHBG-10
- Seroquel Group (Experimental): Subjects who are on a stable dose of Seroquel and taking 500 mg of IHBG-10 15 minutes before the three main meals of the day.
  Interventions: Dietary Supplement: IHBG-10
- Zyprexa Group (Experimental): Subjects who are on a stable dose of Zyprexa and taking 500 mg of IHBG-10 15 minutes prior to the three main meals of the day.
  Interventions: Dietary Supplement: IHBG-10

INTERVENTIONS:
Other: Placebo — Placebo
  Other Names: sugar pill
  Arms: Control Group
Dietary Supplement: IHBG-10 — 500 mg IHBG-10
  Other Names: IHBG10
  Arms: Risperdal Group; Seroquel Group; Zyprexa Group

SUMMARY:
This is a pilot study to determine the safety and efficacy of an investigational product (IHBG-10) on weight change and changes in body composition in subjects who have been taking a stable dose of certain anti-psychotic medications for longer than three months.

DETAILED DESCRIPTION:
A total of 80 subjects will be enrolled in this study: 20 subjects will be randomized to receive placebo, and 60 will be randomized to receive the investigational product (20 who are on a stable dose of Seroquel, 20 who are on a stable dose of Risperdal, and 20 who are on a stable dose of Zyprexa). The investigational product or placebo will be taken 15 minutes prior to the three main meals of the day. Subjects will continue to take their prescribed anti-psychotic medications. Participation in this study involves four study visits.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 18 and older
* Agree to keep diet, exercise and all current health habits stable during participation in the study
* Currently on a stable dose of Risperdal (Risperidone), Seroquel (Quetiapine) and/or Zyprexa (Olanzapine) for at least three months

Exclusion Criteria:

* Current active acute psychotic episode
* Women who are pregnant, breastfeeding, or planning to become pregnant
* Prior bariatric surgery
* Use of prescription or over-the-counter appetite suppressants, herbal products or other medications for weight loss within the past month
* Obesity as a result of a clinically-diagnosed endocrine problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Weight | 12 weeks

SECONDARY OUTCOMES:
Body composition | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Edward Zawada, MD, Principal Investigator — Avera McKennan Hospital & University Health Center
Locations (1):
- Avera Research Institute, Sioux Falls, South Dakota, United States